CLINICAL TRIAL: NCT01216774
Title: The Role of Mechanical Stress and Muscle Fatigue in Strength Gains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: S52680
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2010-09

CONDITIONS: Strength Training; Muscle Strength, Muscle Mass, Inflammatory Processes
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Low load + fatigue (Experimental)
  Interventions: Other: Strength training
- High load (Active Comparator)
  Interventions: Other: Strength training
- Low load (Placebo Comparator)
  Interventions: Other: Strength training

INTERVENTIONS:
Other: Strength training — Leg extension exercise:
  Experimental: 60 repetitions at 20-25% of 1RM, 10-12 repetitions at 40% of 1RM Active Comparator: 10-12 repetitions at 80% of 1RM Placebo Comparator: 10-12 repetitions at 40% of 1RM

SUMMARY:
The purpose of this study is to compare the impact of different levels of mechanical stress and muscle fatigue in strength training conditions on muscle strength, muscle mass and inflammatory processes.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Knee pathology
* Systematic training

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Force-velocity characteristics of knee extensors with biodex dynamometer | Pre and post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Kinesiology and Rehabilitation Sciences, Leuven, Leuven, Belgium